CLINICAL TRIAL: NCT06226467
Title: Neurobehavioral Affective Control Training (N-ACT): A Randomized Waitlist-controlled Pilot Trial to Evaluate a Novel Cognitive Remediation Program for Emotion-related Impulsivity and Rumination
Brief Title: Neurobehavioral Affective Control Training
Acronym: N-ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of Bergen (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01-15949
Record Dates: First submitted 2023-11-06; First posted 2024-01-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Emotional Distress; Impulsive Behavior; Mood Lability; Mood Instability; Rumination; Psychopathology; Affective Symptoms
Keywords: Cognitive Control; Cognitive Training; Emotion Regulation; Emotional Response Inhibition; Emotional Working Memory; Executive Functioning; Urgency; Self-regulation; Cognitive Remediation
MeSH Terms: conditions — Impulsive Behavior; Rumination Syndrome; Affective Symptoms; Emotional Regulation; Self-Control

STUDY DESIGN:
Intervention Model Description: Randomized waitlist-controlled trial or randomized delayed intervention-controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-ACT without delay (Experimental): After a baseline in-person assessment session (Week 1), participants randomly assigned to the experimental condition (i.e., "N-ACT without delay") will complete one week of pre-intervention ecological momentary assessment (EMA; Week 2), then the intervention (Weeks 3-10), followed by a post-treatment in-person assessment session with comparable measures to baseline (Week 11) and a second week of (post-intervention) EMA (Week 12).
  Interventions: Behavioral: Neurobehavioral Affective Control Training
- Waitlist control (Other): Participants randomly assigned to the two-month waitlist control condition will be recontacted approximately 10 weeks after the baseline in-person assessment session (Week 1) to complete a second assessment session (with comparable measures) post-waitlist, prior to starting the N-ACT program. The post-waitlist assessment session (Week 11) after the waitlist period (Weeks 2-10) will precede a series of procedures equivalent to the experimental ("N-ACT without delay") arm: One subsequent week of pre-intervention (post-waitlist) ecological momentary assessment (EMA; Week 12), then eight weeks of N-ACT (Weeks 13-20), followed by a third and final in-person (post-intervention) assessment (Week 21) with parallel procedures to the baseline and post-waitlist sessions, as well as a second week of EMA (Week 22). All study procedures are identical between the two trial arms, with the exception of an added eight-week waitlist and post-waitlist assessment for participants in the control condition.
  Interventions: Behavioral: Neurobehavioral Affective Control Training

INTERVENTIONS:
Behavioral: Neurobehavioral Affective Control Training — The N-ACT program comprises a series of eight training sessions, lasting one hour each, over two months. N-ACT sessions will be guided by a cognitive training "coach" (supervised by a licensed mental health clinician), who will explain intervention procedures and rationale, offer relevant psychoeducation, and use motivational interviewing principles to provide encouragement and support. In addition to coach-led content, participants will spend about half of each weekly training session (~30 minutes) practicing two computer-based adaptive training tasks targeting affective control.
  Other Names: N-ACT

SUMMARY:
The goal of this clinical trial is to test a new cognitive training program to improve emotion regulation in adults. The investigators' primary aim is to determine whether participating in this program addresses two key features of emotion dysregulation associated with psychiatric disorders: (1) emotion-related impulsivity and (2) rumination. The investigators will further evaluate participants' perceived acceptability and feasibility of treatment procedures. Secondarily, the investigators will examine the effects of this cognitive training intervention on psychiatric symptoms and overall functioning. The researchers will compare the cognitive training program to a waitlist control.

Participants will be asked to complete eight weekly sessions (over two months) involving cognitive training exercises with a "coach", in addition to a baseline assessment before starting the intervention and post-treatment assessment. Each assessment includes a combination of in-person and remote data collection using self-report questionnaires, psychophysiology, and a neuropsychological battery. Participants will also complete one week of ecological momentary assessment before and after the intervention as well as a set of follow-up questionnaires administered remotely six weeks following their final training session. Researchers will compare participants randomly assigned to complete the intervention without delay to a control group of participants randomly assigned to a two-month waitlist before joining the intervention. Before beginning cognitive training, participants in the control condition will complete an additional pre-intervention/post-waitlist assessment, which will follow parallel procedures to the initial baseline assessment.

DETAILED DESCRIPTION:
This randomized waitlist-controlled pilot trial will enroll adult participants who self-report high levels of rumination and/or emotion-related impulsivity. The primary aim of this study is to examine the acceptability, efficacy, and feasibility of Neurobehavioral Affective Control Training (N-ACT) as a novel therapeutic approach to reduce emotion-related impulsivity and rumination in adults by improving two types of affective inhibitory control: (1) emotional response inhibition and (2) emotional working memory. Secondarily, study investigators will test anticipated transfer effects of N-ACT on other behavioral indices of cognitive control (beyond emotional response inhibition and emotional working memory) and other subjective measures of emotion dysregulation (beyond trait emotion-related impulsivity and rumination), as well as on psychopathology symptom severity and functional impairment. In addition to performing intent-to-treat analyses, the investigators will conduct analyses to evaluate the extent to which program adherence predicts hypothesized intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Current residency in the state of California
* Elevated levels of rumination and/or emotion-related impulsivity

Exclusion Criteria:

* Insufficient English language literacy to understand study procedures (as assessed by self-report)
* Careless or inattentive responding as indicated by (a) failing 50% or more of "attention check" items embedded in the online screening questionnaires, (b) overly rapid responding (i.e., mean response time of less than two seconds for multiple choice items), or (c) qualitative review of long strings of identical entries on screening/baseline questionnaire items that suggest data invalidity
* Positive history of brain tumors, neurological disorders, or head injuries (with loss of consciousness more than five minutes and/or more than two separate instances of clinically-significant head trauma)
* Recent (i.e., past three months) alcohol/other substance use disorders or current psychosis (as assessed by the Mini International Neuropsychiatric Interview; MINI)
* Active suicidal ideation paired with either (1) plan and/or intent or (2) lifetime history of suicide attempts (as assessed by the Columbia Suicide Severity Rating Scale; C-SSRS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Emotion-related impulsivity (ERI) | (T1) Baseline (Week 1); (T2) Post-waitlist or post-intervention (Week 11)
  ERI will be measured using the self-rated Three-Factor Impulsivity Index "Feelings Trigger Action" scale using standard scoring methods (range: 1-5; larger values indicate higher levels of this characteristic). The researchers will perform a 2 (Arm/Condition: Experimental vs. Control) X 2 (Time: T1 vs. T2) Multivariate Analysis of Covariance (MANCOVA) to evaluate if N-ACT completion is associated with greater pre/post reductions in ERI scores compared to waitlist, as predicted.
Rumination | (T1) Baseline (Week 1); (T2) Post-waitlist or post-intervention (Week 11)
  Rumination will be measured using the self-rated "Brooding" subscale of the Ruminative Responses Scale using standard scoring methods (range: 5-20; larger values indicate higher levels of this characteristic). The researchers will perform a 2 (Arm/Condition: Experimental vs. Control) X 2 (Time: T1 vs. T2) MANCOVA to evaluate if N-ACT completion is associated with greater pre/post reductions in Rumination scores compared to waitlist, as predicted.

SECONDARY OUTCOMES:
Emotional Response Inhibition | (T1) Baseline (Week 1); (T2) Post-waitlist or post-intervention (Week 11)
  Valence-specific indices of stop-signal reaction time (SSRT) will be derived from the Emotional Stop-Signal Task using standard scoring procedures (measured in milliseconds, with larger values indicating less efficient emotional response inhibition, i.e., longer latency of relevant inhibitory processing). The researchers will perform a 2 (Arm/Condition: Experimental vs. Control) X 2 (Time: T1 vs. T2) MANCOVA to evaluate if N-ACT completion is associated with greater pre/post improvement in emotional response inhibition across valence (i.e., reductions in Positive SSRT and Negative SSRT, tested in the same model) compared to waitlist, as predicted, suggesting improvement in targeted aspects of affective control.
Emotional Working Memory | (T1) Baseline (Week 1); (T2) Post-waitlist or post-intervention (Week 11)
  Valence-specific indices of working memory accuracy will be derived from the Memory and Affective Flexibility Task using standard scoring procedures (range: 0.00%-100%, measured as a percentage of working memory trials with correct responses over the total number of trials within each stimulus valence category, with larger values indicating more accurate working memory recall). The researchers will perform a 2 (Arm/Condition: Experimental vs. Control) X 2 (Time: T1 vs. T2) MANCOVA to evaluate if N-ACT completion is associated with greater pre/post improvement in emotional working memory across valence (i.e., increases in Positive Working Memory Accuracy and Negative Working Memory Accuracy, tested in the same model) compared to waitlist, as predicted, suggesting improvement in targeted aspects of affective control.
Affective Flexibility | (T1) Baseline (Week 1); (T2) Post-waitlist or post-intervention (Week 11)
  Valence-specific indices of accuracy (range: 0.00%-100%, measured as a percentage of "switch" trials with correct responses over the total number of trials within each stimulus valence category, with larger values indicating more accurate affective stimulus processing) and reaction time (RT; measured in milliseconds, with larger values indicating less efficient affective flexibility, i.e., longer latency of stimulus processing) will be derived from the Memory and Affective Flexibility Task using standard scoring procedures. A 2 (Arm/Condition: Experimental vs. Control) X 2 (Time: T1 vs. T2) MANCOVA will be used to evaluate if N-ACT completion is associated with greater pre/post improvement in affective flexibility across valence (i.e., increases in Accuracy and decreases in RT for Positive and Negative stimuli, tested in the same model) compared to waitlist, as predicted, suggesting near-transfer of trained abilities to non-targeted aspects of affective control.
Cold Response Inhibition | (T1) Baseline (Week 1); (T2) Post-waitlist or post-intervention (Week 11)
  Stop-signal reaction time (SSRT) will also be derived from the traditional (i.e., non-emotional) version of the Stop-Signal Task using standard scoring procedures (measured in milliseconds, with larger values indicating less efficient cold response inhibition, i.e., longer latency of relevant inhibitory processing). A 2 (Arm/Condition: Experimental vs. Control) X 2 (Time: T1 vs. T2) MANCOVA will be used to evaluate if N-ACT completion is associated with greater pre/post improvement in cold response inhibition (i.e., reductions in SSRT) compared to waitlist, as predicted, suggesting far-transfer of trained abilities to non-targeted aspects of cold cognitive control.
Cold Working Memory | (T1) Baseline (Week 1); (T2) Post-waitlist or post-intervention (Week 11)
  Cold working memory performance will be derived from the Backwards Digit Span task using standard scoring procedures (measured as mean digit span, i.e., the average number of correctly-recalled digits in reverse order from their presentation, with larger values indicating better cold working memory updating capacity). A 2 (Arm/Condition: Experimental vs. Control) X 2 (Time: T1 vs. T2) MANCOVA will be used to evaluate if N-ACT completion is associated with greater pre/post improvement in cold working memory (i.e., increases in mean digit span) compared to waitlist, as predicted, suggesting suggesting far-transfer of trained abilities to non-targeted aspects of cold cognitive control.
Internalizing factor score | (T1) Baseline (Week 1); (T2) Post-intervention (Week 11 or Week 21 for control arm)
  Internalizing psychopathology will be represented as a latent variable derived from raw scores on the self-rated (range: 1-5) Inventory of Depression and Anxiety Symptoms (IDAS) using confirmatory factor analysis (CFA), which is expected to produce a single-factor solution. CFA will be used to generate aggregated, standardized Z-scores on a latent composite "Internalizing" variable at each assessment point (coded such that larger values reflect greater symptom severity). Structural equation modeling of measurement invariance (between groups and within-subjects over time) will test hypothesized treatment effects on Internalizing psychopathology as a latent construct, which is expected to decrease in magnitude from pre- (T1) to post-intervention (T2).
Externalizing factor score | (T1) Baseline (Week 1); (T2) Post-intervention (Week 11 or Week 21 for control arm)
  Externalizing psychopathology will be represented as a latent variable derived from raw scores on self-rated scales pertaining to substance use (range: 1-5) from the revised Externalizing Symptom Inventory using confirmatory factor analysis (CFA), which is expected to produce a single-factor solution. CFA will be used to generate aggregated, standardized Z-scores on a latent composite "Externalizing" variable at each assessment point (coded such that larger values reflect greater symptom severity). Structural equation modeling of measurement invariance (between groups and within-subjects over time) will test hypothesized treatment effects on substance-related Externalizing psychopathology as a latent construct, which is expected to decrease in magnitude from pre- (T1) to post-intervention (T2).

OTHER OUTCOMES:
Acceptability | Final (i.e., eighth) N-ACT training session (Week 10 or Week 20 for control arm)
  Mean scores on the "Interest/Enjoyment" subscale of the Adapted Intrinsic Motivation Inventory will be used to evaluate the perceived acceptability of the N-ACT program. This self-report index comprises an average of seven items each rated on a 7-point Likert scale (range: 7-49), with larger values indicating greater subjective levels of treatment acceptability. Participants will complete these items during the final intervention session. An average rating of 35 (out of 49) points on this scale will be used as a quantitative "cutoff" score indicating hypothesized adequacy of the intervention's acceptability.
Adherence | Final (i.e., eighth) N-ACT training session (Week 10 or Week 20 for control arm)
  Adherence for each participant will be calculated as a function of (1) number of completed N-ACT training task trials divided by the total number of trials, i.e., individual differences in "dosage" of training and (2) attendance rates over the eight weekly N-ACT training sessions (range: 0.00%-100%, measured as percentages, with larger values reflecting higher levels of treatment adherence and feasibility). Median person-level adherence levels are expected to be between 70-75%, and are expected to decrease at the group-level by approximately 5% each week, with the majority of participants (i.e., > 66%) attending and completing all eight N-ACT training sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Sheri L. Johnson, Ph.D., Principal Investigator — University of California, Berkeley; J.D. Allen, Ph.D., Study Director — University of California, Berkeley; Åsa Hammar, Ph.D., Study Director — University of Bergen
Locations (1):
- University of California, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Measures, data, and analysis scripts will be shared through an Open Science Framework (OSF) registration.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will be shared within one year after data collection ends and available for seven years.
Access Criteria: Data will be made available to the public through OSF.

REFERENCES:
- [Derived] Allen KJD, Elliott MV, Ronold EH, Mason L, Rajgopal N, Hammar A, Johnson SL. Cognitive Training for Emotion-Related Impulsivity and Rumination: Protocol for a Pilot Randomized Waitlist-Controlled Trial. JMIR Res Protoc. 2025 Feb 19;14:e54221. doi: 10.2196/54221. PMID 39970439